CLINICAL TRIAL: NCT05279248
Title: Immunogenicity and Safety of Concomitant Inoculation of Recombinant Human Papillomavirus Bivalent (Types 16,18) Vaccine (Escherichia Coli) and Measles Mumps and Rubella Combined Vaccine, Live
Brief Title: The Immunogenicity and Safety of the Vaccination of Human Papillomavirus Vaccine and Measles-Mumps-Rubella Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZJCDC202102801
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Human Papilloma Virus Infection Type 16; Human Papilloma Virus Infection Type 18; Measles; Rubella; Mumps
Keywords: Immunogenicity; Safety; Recombinant Human Papillomavirus Bivalent (Types 16,18) Vaccine (Escherichia coli); Measles Mumps and Rubella Combined Vaccine, Live
MeSH Terms: conditions — Measles; Rubella; Mumps; Escherichia coli Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Participants in this arm will be simultaneously administrated with one dose of HPV 16/18 bivalent vaccine and one dose of MMR vaccine. six month later, they are going to receive a second dose of HPV 16/18 bivalent vaccine.
  Interventions: Biological: HPV+MMR（0d），HPV（6m）
- Group B (Active Comparator): Participants in this arm will be receieve HPV 16/18 bivalent vaccine according to 2-dose schedule (0,6 months) first. After finished HPV vaccination, they are going to receive MMR vaccine at the 7th month.
  Interventions: Biological: HPV（0d），HPV（6m），MMR（7m）
- Group C (Active Comparator): Participants in this arm will be receieve MMR vaccine first. One month later, they are going to receieve HPV 16/18 bivalent vaccine according to 2-dose schedule (1,7 months)
  Interventions: Biological: MMR（0d），HPV（1m），HPV（7m）

INTERVENTIONS:
Biological: HPV+MMR（0d），HPV（6m） — Simultaneously administrated with MMR vaccine and HPV 16/18 bivalent vaccine at first. And six months later, administrated with the second dose of HPV 16/18 bivalent vaccine.
  Arms: Group A
Biological: HPV（0d），HPV（6m），MMR（7m） — Administrated with HPV 16/18 bivalent vaccine according to 2-dose schedule (0,6 months).And at the 7th month , administrated with MMR vaccine.
  Arms: Group B
Biological: MMR（0d），HPV（1m），HPV（7m） — Administrated with MMR vaccine at first day. And administrated with HPV 16/18 bivalent vaccine according to 2-dose schedule (1,7 months).
  Arms: Group C

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of Recombinant Human Papillomavirus Bivalent (Types 16,18) Vaccine (Escherichia coli) （HPV）and Measles Mumps and Rubella Combined Vaccine, Live（MMR）

DETAILED DESCRIPTION:
Main subjects:

To evaluate the immunogenicity of HPV vaccine and MMR vaccine at the same time but at different sites as not inferior to vaccination of HPV vaccine or MMR vaccine alone.

Secondary subjects:

To evaluate the safety of simultaneous administration of HPV vaccine and MMR vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged between 13 and 14 years when they receive the first vaccination (13≤age<15);
2. Participants aged 13-14 years whose legal guardian can provide identity certificate, or representative can provide authorization;
3. Judged as healthy and eligible for vaccination by the investigators through a self-reported medical history and some physical examinations;
4. Participants aged 13-14 years, able to sign or whose legal guardian agree to sign the written informed consent; or participants aged 18-26 years and agree to sign the written informed consent;
5. Able to comply with the requests of the study;
6. Axillary temperature not higher than 37.0°C; Nonpregnancy verified by a urine pregnancy test;

Exclusion Criteria:

1. Pregnant or lactating woman and any woman who are willing or intend to become pregnant in next 7 months;
2. Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the first vaccination, or plan to use during the study period;
3. Participants who received an immunosuppressive agent or other immunomodulator agent for a long term (for 14 days or more) within 6 months of the first vaccination, or systematic corticosteroid (however, a topical corticosteroid is allowed, such as ointment, eye drops, inhalant, or nasal spray);
4. Participants who received immunoglobulin and/or blood product 3 months prior to the first vaccination, or planned to receive during the study period;
5. Use of any inactivated vaccine 14 days preceding dosing of study vaccine or attenuated vaccine 21 days before the enrollment;
6. Participants had fever (auxiliary temperature ≥38.0 °C) within 3 days prior to vaccination, or any acute disease requiring systematic antibiotics or antiviral therapy within the past 5 days;
7. Concurrently participating another clinical trial;
8. Participants who have received HPV vaccines;
9. Participants with immunodeficiency disease (such as HIV positive), primary disease in vital organs, cancer (or precancerous lesion), or chronic history of immunological disease requiring treatment (including systemic lupus erythematosus), rheumatoid arthritis, asplenia or splenectomy due to any conditions, and other immunological diseases that may impact immune response as considered by investigator), etc.;
10. Participants with a history of allergy, including severe adverse reactions due to the past vaccination, such as hypersensitivity, urticaria, dyspnea, angioneurotic edema, or abdominal pain;
11. Participants with asthma, which is unstable in the past 2 years, requiring emergency treatment, hospitalization, or oral or intravenous corticosteroid;
12. Participants with concurrent severe medical disorders, such as hypertension, heart disease, diabetes mellitus, or hyperthyroidism, etc.;
13. Participants with coagulation dysfunction (such as coagulation factor deficiency, blood-clotting disorder, or platelet disorder) or coagulation disorders, as diagnosed by a physician;
14. Participants with epilepsy, excluding febrile epilepsy in patients under 2 years old, alcoholic epilepsy 3 years prior to alcohol abstinence, or pure epilepsy requiring no treatment within the past 3 years;
15. Participants who are not compliant to the study's requirements due to psychological conditions, or those with prior or existing mental disease or bipolar psychosis which are not well controlled within the past 2 years and require taking drugs, or those with suicidal tendency within the past 5 years;
16. According to the investigator's judgment, there might be some medical, psychological, social or occupational factors which might impact on the individual to obey the protocol or sign the informed consent;

Ages: 13 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate the seroconversion rates and geometric mean concentrations of anti-HPV 16 and 18 at Months 7 (type specific neutralizing antibody) | Specific neutralizing antibodies at 7 months after first dose
  Detect the level of anti-HPV 16 and 18 specific neutralizing antibodies at one month after the second dose to determine whether group A is non-inferior to group B
Evaluate seroconversion rates and geometric mean concentrations of anti-measles at the 1st month after MMR vaccination | 1 months after vaccination
  Detect the level of anti-measles specific neutralizing antibodies at one month after MMR vaccination to determine whether group A is non-inferior to group C
Evaluate seroconversion rates and geometric mean concentrations of anti-rubella at the 1st month after MMR vaccination | 1 months after vaccination
  Detect the level of anti-rubella specific neutralizing antibodies at one month after MMR vaccination to determine whether group A is non-inferior to group C
Evaluate seroconversion rates and geometric mean concentrations of anti-mumps at the 1st month after MMR vaccination | 1 months after vaccination
  Detect the level of anti-mumps specific neutralizing antibodies at one month after MMR vaccination to determine whether group A is non-inferior to group C

SECONDARY OUTCOMES:
Local and systematic adverse events/reactions occurred within 7 days after each vaccination | During the 7-day (Day 0-6) period following each vaccination
  Adverse reactions associated with vaccine will be observed in subjects after vaccination. To evaluate number of adverse events/reactions compared with non-simultane vaccination group.
Adverse events/reactions occurred within 30 days after each vaccination | Within 30 days (Day 0-30) after any vaccination
  To evaluate number of adverse events/reactions compared with non-simultane vaccination group.
Serious adverse events occurred throughout the study | Up to 7 months
  safety analysis. To evaluate number of SAEs compared with the non-simultane vaccination group.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Yuecheng Center for Disease Control and Prevention, Shaoxing, Zhejiang
  - Wuyi Center for Disease Control and Prevention, Wuyi, Zhejiang

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263